CLINICAL TRIAL: NCT01710878
Title: Multicenter Clinical Study Assessing the Performance and the Safety of the Second Generation Antimicrobial Graft in Abdominal Position
Brief Title: Performance and Safety of a Second Generation Antimicrobial Graft in Abdominal Position
Acronym: SYNERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR07-001
Record Dates: First submitted 2012-10-10; First posted 2012-10-19 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Abdominal Aorta Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intergard Synergy Graft (Other)
  Interventions: Device: Intergard Synergy Graft

INTERVENTIONS:
Device: Intergard Synergy Graft

SUMMARY:
Safety and performance of an anti-microbial vascular graft in the treatment of aneurysmal and occlusive disease of the abdominal aorta.

DETAILED DESCRIPTION:
The purpose of this multi center, single arm study is to demonstrate the safety and performance of the Second Generation Anti-Microbial (InterGard Synergy) vascular graft in the treatment of aneurismal and occlusive diseases of the abdominal aorta.

The primary endpoint is the assessment of primary and secondary graft patency. The secondary endpoints were the assessment of adverse events and the assessment of triclosan and silver contents in the serum over the time.

ELIGIBILITY:
Inclusion Criteria:

Patient aged 18-85 years

Patient presenting with an aorto-iliac occlusion (obstruction of flow) or stenosis, or aorto-iliac aneurysm and eligible for a revascularization with a bifurcated graft

Exclusion Criteria:

Patient treated as an emergency

Patient included in another investigation

Patient pregnant or lactating or woman of childbearing potential

Patient with a known allergy to the material device used (collagen, triclosan, silver)

Patient with previous aorto-iliac bypass or replacement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary Graft Patency | Up to 36 months
  Defined as uniterrupted flow with no interventions. Follow-up timeframes - 1, 6, 12, 24, and 36 months

SECONDARY OUTCOMES:
Secondary endpoint - assessment of AEs | Up to 36 months
  Follow-up timeframes - 1, 6, 12, 24, and 36 months

OTHER OUTCOMES:
Secondary endpoint - levels of silver and triclosan | Up to 30 days
  Serum levels prior to surgery, 1 day post-implant, discharge and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Ricco, MD, Principal Investigator — CHU La Milétrie
Locations (8):
- France (7):
  - CHRU, Angers
  - CHU Jean Minjoz, Besançon
  - CHU Dupuytren, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Hôpital G. et R. Laennec, Nantes
  - Hôpital Pompidou, Paris
  - CHU La Milétrie, Poitiers
- Krankenhaus Nordwest, Frankfurt, Germany